CLINICAL TRIAL: NCT06070428
Title: ACHIEVE GREATER: Addressing Cardiometabolic Health In Populations Through Early Prevention in the GREAT LakEs Region Project 4: Portable Air Cleaners to Treat Heart Failure and Negate Disparities of Environment and Race (PATHFINDER)
Brief Title: Project 4: ACHIEVE PATHFINDER
Acronym: PATHFINDER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Wayne State University (Other)
Responsible Party: Principal Investigator, David Lanfear, Senior Staff Physician, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16658
Record Dates: First submitted 2023-09-26; First posted 2023-10-06 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
Keywords: Health Disparities; Portable Air Cleaner; Exposure; Air Pollution
MeSH Terms: conditions — Heart Failure | interventions — Chromosomes, Artificial, P1 Bacteriophage; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: ACHIEVE-P4: PATHFINDER is a randomized, blinded clinical trial of portable air cleaners (PAC) provided at the time of hospital discharge to Heart Failure (HF) patients. It will be carried out at Henry Ford Hospitals.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators will use mixed block sizes (2, 4, 6) for randomizing participants. Control versus PAC interventional units will be prepared by study staff who will not directly enroll patients. The crosswalk for patient study ID and randomization status will be kept in a secure separate location so that PI and staff in charge of data analysis will not be aware of randomization status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PAC Intervention Arm (Active Comparator): Participants randomized to the interventional arm will be given 2 PAC units with HEPA filters inside to be used in the home: one in the room patient sleeps in, the other in the living area of the home. Participants will also be given an air quality monitor. Study staff will educate the patient on use of the filters and monitor.
  Patients will be seen in clinic for 30-day and 90-day follow-up visits. Blood pressure, blood draw for biomarker levels, 6-minute walk distance, and questionnaires will be completed.
  Patients will be allowed to keep the PAC at the end of the trial and will be informed at that time how to purchase additional filters.
  Interventions: Other: PAC provision at hospital discharge
- Control non-interventional Arm (Sham Comparator): Participants randomized to the non-interventional arm will be given 2 PAC units without HEPA filters inside to be used in the home: one in the room patient sleeps in, the other in the living area of the home. Participants will also be given an air quality monitor. Study staff will educate the patient on use of the filters and monitor.
  Patients will be seen in clinic for 30-day and 90-day follow-up visits. Blood pressure, blood draw for biomarker levels, 6-minute walk distance, and questionnaires will be completed.
  Patients will be allowed to keep the PAC at the end of the trial and will be informed at that time how to purchase additional filters.
  Interventions: Other: Control non-intervention; PAC without filter

INTERVENTIONS:
Other: PAC provision at hospital discharge — Patients randomized to receive the intervention will receive two PACs fitted with True HEPA filters.
  Other Names: Portable Air Cleaner HEPA Filter
  Arms: PAC Intervention Arm
Other: Control non-intervention; PAC without filter — Patients randomized to the control non-interventional arm will receive two PACs with no filters inserted.
  Other Names: PAC with Sham
  Arms: Control non-interventional Arm

SUMMARY:
ACHIEVE-P4: PATHFINDER is a randomized, blinded clinical trial of portable air cleaners (PAC) provided at the time of hospital discharge to Heart Failure (HF) patients. It will be carried out at Henry Ford Hospitals. This project is part of the ACHIEVE GREATER (Addressing Cardiometabolic Health In Populations Through Early PreVEntion in the GREAT LakEs Region) Center (IRB 100221MP2A). The ACHIEVE GREATER Center involves several separate but related projects that aim to prolong lifespan among Detroit, MI and Cleveland, OH, for three chronic conditions, hypertension (HTN, Project 1), heart failure (HF, Projects 2 & 4) and coronary heart disease (CHD, Project 3). The present study is Project 4 (Aim 1) a randomized clinical trial titled: Portable Air cleaners to Treat Heart Failure and Negate Disparities of Environment and Race (PATHFINDER), of the ACHIEVE GREATER Center.

Project 4 is a randomized, double-blind, parallel limb trial of 400 patients with hospitalized HF who will be provided active PAC vs sham at discharge from HFH.

Participants will receive two PACs at discharge and an indoor PM2.5 sensor. PACs will be randomized to either active PAC with HEPA filters or sham PAC without HEPA filters.

Researchers will compare the following outcomes of the two groups (more outcomes below in Outcome Measures section):

1. Change in NTproBNP from baseline to 90 days
2. Home PM2.5 levels from baseline to 90 days
3. Clinical events such as death and hospitalization will be monitored

DETAILED DESCRIPTION:
Project 4 of ACHIEVE GREATER aims to improve outcomes for symptomatic (Stage C) HF. This is vitally important because HF is the most common final manifestation of cardiometabolic diseases in the U.S., accounting for nearly 400,000 deaths and 900,000 hospitalizations per year. Growing evidence implicates air pollutants adversely impact HF and its prognosis. For example, among 12,474 HF patients in North Carolina, hospital readmission rates at 90-days were increased by 13-14% for every 1 μg/m3 elevation in fine particulate matter <2.5 µm air pollution (PM2.5) levels. While average U.S. air quality has improved, urban communities continue to have higher levels of exposure. Indeed, Detroit residents face the highest PM2.5 concentrations in Michigan (97th percentile for the U.S.). We hypothesize that this may contribute to worse outcomes among HF patients in Detroit, including an unacceptably high rate of death or rehospitalization (22% based on Henry Ford Health [HFH] data for 2022) at 90-days post-discharge. To combat this problem, we propose to test an emerging therapeutic intervention, the portable air cleaner (PAC), that we hypothesize will reduce personal-level exposure to PM2.5 resulting in improved clinical outcomes for HF patients. This novel intervention is both practical and scalable, and thus has the potential to revolutionize the treatment of HF and improve related outcomes nationwide.

ELIGIBILITY:
Inclusion Criteria:

1. Currently in the emergency room or hospitalized with plan to be discharged to home, or
2. Diagnosis of heart failure
3. BNP>200 ng/L or NTproBNP>1000 ng/L during hospitalization or within 1 month prior to screening
4. Expected ability to fully participate in study (can tolerate study processes, no long travel)

Exclusion Criteria:

1. Hemodialysis dependent
2. If dialysis is being considered by participant's care team and their eGFR value is <30 mL/min/1.73 sq m
3. Life expectancy of less than one year
4. Inability to provide written informed consent
5. Age less than 18 years old
6. Patients with a left ventricular assist device (LVAD)
7. Heart transplant recipients
8. Individuals who regularly use a HEPA air cleaner in their home at screening
9. Current smokers of nicotine or marijuana
10. Severe aortic or mitral valve disease
11. Has a scheduled, non-diagnostic cardiac procedure within 30 days prior, or in the next 90 days from screening (e.g. PCI, resynchronization, any cardiac surgery)
12. If the PI decides for any reason that participation in the trial is not in the best interest of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The impact of PAC use for 90 days after hospital discharge for HF compared to sham on NTproBNP level. | Baseline at hospital discharge to 90 days.
  Change in NTproBNP from baseline to 90 days. This will be determined by comparing the NTproBNP value at the 90-day follow up visit versus the baseline NTproBNP value measured from blood draw at enrollment/randomization visit (within 48 hours of hospital discharge).

SECONDARY OUTCOMES:
The effect of PAC use on home PM2.5 levels in active PAC group versus sham group | Baseline to 90 days
  Each participant will be provided an indoor PM2.5 sensor to measure in-home PM2.5 levels
The effect of PAC use on clinical events (death) in the active PAC group versus sham group | Baseline to 90 days
  Clinical events such as death will be monitored primarily by EMR data.
The effect of PAC use on clinical events (hospitalization) in the active PAC group versus sham group | Baseline to 90 days
  Clinical events will be monitored primarily by EMR data, but patients will also be queried at study visits regarding hospitalization.

OTHER OUTCOMES:
Impact of PAC on hsCRP | 30 and 90 days post-enrollment
  hsCRP and hsTroponin will be measured at 30 and 90 days post-enrollment
Impact of PAC use on health status | Baseline, 30 and 90 days post enrollment
  Change in health status will be evaluated by use of the Kansas City Cardiomyopathy Questionnaire (KCCQ) a validated health status tool for detecting clinically important changes. The score will be represented on a 0-to-100 scale; lower scores represent more severe symptoms and scores of 100 represent no limitations.
Impact of PAC on hsTroponin | 30 and 90 days post-enrollment
  hsTroponin will be measured at 30 and 90 days post-enrollment

CONTACTS AND LOCATIONS:
Overall Officials: David Lanfear, MD, Principal Investigator — Henry Ford Health
Locations (1):
- Henry Ford Health, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No